CLINICAL TRIAL: NCT03746964
Title: Prospective Evaluation of the Biomechanical Properties of the Thoracic Aorta Coupling Magnetic Resonance Imaging and In-vitro Elasticity Tests in Patients With Ascending Aortic Aneurysm
Acronym: MECATHOR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MORGANT 2018 MECATHOR
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Patient With Ascending Aortic Aneurysm With Surgical Indication for Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac MRI — Preoperative cardiac MRI
Other: in-vitro elasticity tests — in-vitro elasticity tests performed on a segment of ascending aorta collected during surgery

SUMMARY:
The biomechanical properties of the aorta are currently poorly understood. A better understanding would optimize surgical indications and monitoring techniques for patients with thoracic aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Patient with ascending aortic aneurysm with surgical indication for replacement
* Age > 18 years old
* Scheduled surgery

Exclusion Criteria:

* Person not affiliated to the national health insurance system
* Protected adult
* Pregnant or breastfeeding woman
* MRI Contraindication
* Emergency surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in preoperative consultation in the cardiovascular and thoracic surgery department.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
aortic compliance by cardiac MRI | Before surgery
In-vitro testing of the elasticity of the aortic wall fragment collected during surgery. | through study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France